CLINICAL TRIAL: NCT07282925
Title: Effects of Cognitive Functional Therapy Versus Kinetic Control Training on Pain, Disability, Movement Control in Patients With Non-specific Low Back Pain
Brief Title: Comparative Effects of Cognitive Functional Therapy With Kinetic Control Training on Non-specific Low Back Pain
Acronym: LBP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Umber Nawaz, Assistant Professor, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/021; U1111-1331-9059 (Registry Identifier: WHO Universal Trial Number)
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain; Non Specific Chronic Low Back Pain
Keywords: Low Back Pain; Non Specific Low Back Pain; Chronic Low Back Pain; Cognitive Functional Therapy; Kinetic Control Training; Pain; Disability; Movement Control
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Functional Therapy (Experimental)
  Interventions: Behavioral: Cognitive Functional Therapy
- Kinetic Control Training (Active Comparator)
  Interventions: Other: Kinetic Control Training

INTERVENTIONS:
Behavioral: Cognitive Functional Therapy — Patients will receive 3 sessions per week for 8 weeks for a total of 24 sessions. Each session will be of 1 hour 15 minutes.
  Standard Physical Therapy will be provided in which patient will receive Hot pack with TENS and perform a set of exercises including Curl up, Bird dog and side bridge back exercises for 5 repetitions.
  Then Cognitive Functional Therapy (CFT) will be applied from day one. CFT is structured into three phases: (1) making sense of pain, (2) exposure with control, and (3) lifestyle changes. Making Sense of Pain : This component reflects the cognitive aspect of Cognitive Functional Therapy. It involves hearing patient's personal narrative about their chronic pain. Exposure with Control: It involves graded exposure to feared movements and functional tasks. Lifestyle Changes: This component focuses on lifestyle factors that contribute to pain and disability. It involves modifying sedentary lifestyle behaviors and encouraging healthy routine.
  Arms: Cognitive Functional Therapy
Other: Kinetic Control Training — Patients will receive 3 sessions per week for 8 weeks. In each session, Standard Physical Therapy will be applied which will be the same in both groups.
  In Kinetic Control Training (KCT), patients will first undergo direction specific movement control tests. These tests will identify direction-specific movement faults (e.g., flexion, extension, rotation control deficits) that contribute to symptoms. Based on these tests, individualized retraining will be provided to the patients. This retraining will improve control of specific muscles which will help reduce pain and improve disability.
  Arms: Kinetic Control Training

SUMMARY:
The goal of this clinical trial is to compare Cognitive Functional Therapy (CFT) with Kinetic Control Training (KCT) in participants with non-specific low back pain. The study wants to see which approach helps lower pain, reduce disability and improve movement control. The main questions it aims to answer is

* Is there difference between Cognitive Functional Therapy and Kinetic control training on pain intensity, disability and movement control in participants with Non Specific Low Back Pain?
* Is there difference between Cognitive Functional Therapy and Kinetic control training on pain catastrophizing and self-efficacy in participants with Non Specific Low Back Pain? Researcher will compare the both CFT and KCT group to see if one treatment is superior to other in treating participants with non-specific back pain.

Participants will

* Attend treatment sessions based on the group they are placed in.
* Take session three times each week for eight weeks.
* They will be asked short questions about their pain, daily activity, and movement throughout the study.

DETAILED DESCRIPTION:
Low back pain (LBP) has the highest prevalence globally among musculoskeletal disorders, affecting around 619 million people in 2020 and it is expected that the number of cases will increase to 843 million by 2050. LBP is defined as the localized pain below the costal margin and above the inferior gluteal folds which may or may not include leg pain. It is commonly categorized as specific and non-specific low back pain. Non-Specific Low Back Pain (NSLBP) accounts for nearly 90% of all cases.

NSLBP is multifactorial and mostly new cases recover within a short time but the condition frequently recurs and may become persistent. An extensive review regarding the management of LBP has stated that exercise plays a fundamental role in treating patients with NSLBP. However, the results regarding the appropriate type of exercise are the subject of controversy. Over the past decades, researchers have advised a variety of exercises. However, despite applying various treatment approaches, conservative treatment for NSLBP yields small effect sizes.

Cognitive Functional Therapy (CFT) is a contemporary exercise intervention developed by Peter O'Sullivan, to address the multidimensional nature of non-specific low back pain. The CFT is structured into three phases: (1) making sense of pain, (2) exposure with control, and (3) lifestyle changes. Rather than adopting a one size fits all approach, CFT provides clinicians with the opportunity to explore the multidimensional nature of NSLBP.

Kinetic Control Training (KCT) developed by Comerford, is a clinical framework focused on the assessment and correction of uncontrolled movement. KCT emphasizes identifying direction-specific movement faults (e.g., flexion, extension, rotation control deficits) that contribute to symptom provocation. KCT utilizes a three-stage retraining process: (1) cognitive facilitation of correct muscle activation; (2) integration into low-load, non-provocative tasks; and (3) progression to complex, functional movements under load and fatigue.

Despite the promising evidence supporting both CFT and KCT, a clear comparative study of their effectiveness in addressing NSLBP is lacking. Most existing studies have focused on one technique or compared it with general exercise. This study seeks to address this gap by evaluating and comparing the effects of Cognitive Functional Therapy and Kinetic Control Training in individuals with NSLBP.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Aged between 19 to 39
* Patients who score 6 points or higher on the Roland-Morris Disability Questionnaire (RMDQ) at the time of screening
* Patients who will have Non-Specific Chronic Low Back pain for at least 3 months duration

Exclusion Criteria:

* If the primary pain area is not the lumbar spine.
* If leg pain is the primary problem.
* If patient have inflammatory disease.
* If patient have progressive neurological disease.
* If patient have red flag disorders (malignancy/cancer, traumas such as fracture).
* Pregnant females.

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Measured by Numeric Pain Rating Scale | It will be measured at baseline, 4 weeks and at 8 weeks.
  Pain intensity will be measured with an 11 point Numeric Pain Rating Scale that is measured from 0 to 10. 0 is no pain, 1-3 indicates mild pain, 4-6 indicates moderate pain and 7-10 is the most severe pain imaginable.
Disability measured by Roland Morris Disability Questionnaire | It will be measured at baseline, 4 weeks and 8 weeks
  Disability will be measured by Roland Morris Disability Questionnaire (RMDQ). The RMDQ is a valid and reliable tool for estimating the level of disability in Low Back Pain patients. It is composed of 24 questions that are to be answered by the patients with answers of either 'Yes' or 'No'. The variation of the total score may range from a score of 0 (no disability) to a score of 24 (maximum disability).
Lumbar Motor Control measured by the Luomajoki Motor Control Test Battery | baseline, 4 week and 8 week
  To evaluate lumbar motor control, the Luomajoki Motor Control Test Battery is employed. This battery includes six individual tests that examine movement control in various positions such as standing, sitting, quadruped, and prone. Each test is scored either 0 or 1, with a total score of 3 or higher indicates impaired motor control

SECONDARY OUTCOMES:
Catastrophizing pain will be measured by Pain Catastrophizing Scale. | baseline, 4 weeks and 8 weeks
  Catastrophizing pain will be measured by 13-item Pain Catastrophizing Scale (PCS). The PCS serves to evaluate catastrophic thinking related to pain. It includes four items rated on a 5-point Likert scale from 0 (not at all) to 4 (all the time), with total scores ranging from 0 to 52.
Self-efficacy will be measured by Pain Self Efficacy Scale | Baseline, 4 weeks and 8 weeks
  Self-efficacy will be measured by Pain Self Efficacy Scale, a 10-item instrument evaluating a patient's confidence in carrying out daily activities despite experiencing pain. Each item is rated on a 7-point scale and higher scores indicate stronger self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Nayab Naseem, Principal Investigator — Lahore University of Biological and Applied Sciences
Locations (2):
- Pakistan (2):
  - Ghurki Trust Teaching Hospital, Lahore, Punjab Province
  - Private Physical Therapy Clinic, Lahore, Punjab Province